CLINICAL TRIAL: NCT06595355
Title: Efficacy and Safety of Intravitreal Injection of Bevacizumab with and Without Oral Curcumin in Diabetic Macular Edema
Brief Title: Efficacy and Safety of Intravitreal Injection of Bevacizumab with and Without Oral Curcumin
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohsen Pourazizi, Dr.Mohsen Pourazizi, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR.ARI.MUI.REC.1402.336
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Macular Edema; Macular Edema; Retinal Neovascularization
Keywords: macular edema; diabetic macular edema; central macular edema; bevacizumab; Diabetic Retinopathy; Retinal Neovascularization
MeSH Terms: conditions — Macular Edema; Retinal Neovascularization; Diabetic Retinopathy | interventions — Bevacizumab; Curcumin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case: Intravitreal injection of bevacizumab with oral curcumin (Experimental): Intravitreal injection of bevacizumab with oral curcumin Inclusion criteria: Patients with center-involving macular edema with macular center thickness of more than 300 microns in OCT 2-Patients who did not receive intravitreal bevacizumab in the last 3 months and intravitreal corticosteroids in the previous 6 months.
  3- The amount of BCVA should not be <20/400. 4-Consent to participate in the study
  Interventions: Drug: bevacizumab with oral curcumin
- Control: Intravitreal injection of bevacizumab with oral placebo (Placebo Comparator): Intravitreal injection of bevacizumab with oral placebo
  Interventions: Drug: bevacizumab with oral placebo

INTERVENTIONS:
Drug: bevacizumab with oral curcumin — According to the recommendation of the American Association of Ophthalmologists, intravitreal injection of bevacizumab with a standard dose of 1.25mg/0.05ml in each group will be performed three times consecutively at one-month intervals. In the simultaneous intervention group, patients will take daily curcumin tablets (sinacurcumin product) at a dose of 40 mg twice a day for three months (at the same time as the start of bevacizumab intravitreal injection treatment).
  Other Names: intervention group
  Arms: Case: Intravitreal injection of bevacizumab with oral curcumin
Drug: bevacizumab with oral placebo — Intravitreal injection of bevacizumab with a standard dose of 1.25mg/0.05ml in each group will be performed three times consecutively at one-month intervals. In the control group, patients will be taking daily placebo tablets twice a day for three months (at the same time as the start of bevacizumab intravitreal injection treatment).
  Other Names: placebo
  Arms: Control: Intravitreal injection of bevacizumab with oral placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of adding curcumin oral treatment to bevacizumab intravitreal injection in patients with central macular edema.

A blind study and a randomized and controlled clinical trial are conducted on diabetic patients with macular edema. The patients are divided into two intervention groups (bevacizumab + curcumin) and control (bevacizumab + placebo).

The evaluation of the central thickness of the macula and the evaluation of the central volume of the macula are the primary goals and the evaluation of the best visual acuity of the patient is the secondary goal.

ELIGIBILITY:
Inclusion Criteria:

Patients with center-involving macular edema with macular center thickness more than 300 microns in OCT 2-Patients who did not receive intravitreal bevacizumab in the last 3 months and intravitreal corticosteroids in the last 6 months.

3- The amount of BCVA should not be <20/400. 4-Consent to participate in the study

Exclusion Criteria:

1. Other retinal diseases except for DME and macular edema due to other causes including uveitis, epiretinal membrane, central retinal vein occlusion, and...
2. Existence of proliferative diabetic retinopathy and patients with a history of vitrectomy
3. Patients with glaucoma, vitreous hemorrhage, age-related macular degeneration (ARMD)
4. Media opacities that limit the interpretation of diagnostic tests
5. Surgery or procedure 3 months before starting treatment
6. Pregnancy or breastfeeding
7. History of allergy to curcumin
8. Use of warfarin
9. Changing the patient's clinical diagnosis or the need for surgical interventions in the course of the disease
10. Change in the patient's general health condition
11. Absence of patient referrals
12. Lack of consent to continue treatment and follow-up

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-09-22 (Estimated)

PRIMARY OUTCOMES:
central macular thickness (CMT) | 3 months
  Changes in central macular thickness (CMT) in patients with oral Curcumin versus patients in the control group
central macular volume (CMV) | 3 months
  Changes in central macular volume (CMV) in patients with oral Curcumin versus patients in the control group

SECONDARY OUTCOMES:
best visual acuity (BCVA) | 3 months
  Changes in best visual acuity (BCVA) in patients with oral Curcumin versus patients in the control group

CONTACTS AND LOCATIONS:
Locations (1):
- Mohsen Pourazizi, Isfahan, Isfahan University of Medical Sciences, Iran

IPD SHARING:
Plan to Share IPD: No